CLINICAL TRIAL: NCT02922790
Title: Feasibility and Smokers' Reactions to DNA Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00075612
Record Dates: First submitted 2016-09-26; First posted 2016-10-04 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Smoking
Keywords: smoker; smoking; cigarette; cessation; DNA; DNA damage; blood draw; feedback; cellular; tobacco; tobacco smoke
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Subjects will review standard health information on the health consequences of smoking.
  Subjects will have blood drawn but it will not be tested for DNA damage.
  Interventions: Behavioral: standard health information
- Biomarker feedback (Active Comparator): Subjects will review this standardized health information, plus receive information on DNA damage along with feedback of their DNA damage.
  Subjects will have blood drawn and the feedback will be presented at Visit 2.
  Interventions: Behavioral: standard health information plus info. on DNA damage
- Biomarker feedback plus (Active Comparator): Subjects will review this standardized health information, information on DNA damage along with feedback of their DNA damage, and will also will see images of their own cells with and without DNA damage.
  Subjects will have blood drawn and the feedback and images will be presented at Visit 2.
  Interventions: Behavioral: Subjects will review standard health information and information on DNA damage, plus pictures of their DNA damage

INTERVENTIONS:
Behavioral: standard health information — Subjects will review standard health information
  Arms: Control
Behavioral: standard health information plus info. on DNA damage — Subjects will review standard health information and information on DNA damage
  Arms: Biomarker feedback
Behavioral: Subjects will review standard health information and information on DNA damage, plus pictures of their DNA damage — Subjects will review standard health information and information on DNA damage, as well as review pictures of their cells' DNA damage
  Arms: Biomarker feedback plus

SUMMARY:
The purpose of the study is to explore how feedback of cellular DNA (Deoxyribonucleic Acid) damage, as a marker of exposure to the genotoxic agents of tobacco smoke, promotes cessation.

DETAILED DESCRIPTION:
The study aims to recruit 50 smokers who are not engaged in quitting. The study will involve two in-person visits. During visit 1, participants will complete a baseline survey and have their blood drawn. Approximately two weeks later, in visit 2, smokers will be randomized in a 1:2:2 ratio to one of three arms:

1. education about harms of smoking (control group);
2. same education plus information on DNA damage and biomarker feedback (biomarker arm) without visual of damage; or
3. same as arm 2 except accompanied with visuals of participants' normal and DNA damage cells. Participants in the this arm will be informed of their proportion of leucocytes showing DNA damage with pictures of their normal and damaged cells.

The goal of the analyses is to obtain effect size estimates (direction, confidence intervals) to inform if results align with hypotheses and obtain insights about reactions about the feedback (Aim 1). The study will collect feasibility data from baseline to three months (e.g., percentage who show up to the sessions, attrition).

ELIGIBILITY:
Inclusion Criteria:

* ages 18+
* smoke > 5 cig/day during the last week
* be open to biomarker feedback
* not actively trying to quit

Exclusion Criteria:

* smoker carbon monoxide level(CO < 10 ppm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Degree of participant understanding of materials, to be measured by a survey | week 3
  Study will measure the extent to which the biomarker information was understood, as measured by a survey
Percentage of subjects who show up to the sessions | Week 1
  Study will collect feasibility data on how many participants come to each visit.
Extent to which participants believe the feedback to be accurate | week 3
  The study will measure the extent to which DNA damage results would be considered accurate using a survey.
Degree of participant understanding of materials, to be measured by an interview | Week 3
  Study will measure the extent to which the biomarker information was understood, as measured by an interview.
Percentage of subjects who show up to the sessions | Week 3
  Study will collect feasibility data on how many participants come to each visit.
Extent to which participants believe the feedback to be trustworthy | Week 3
  The study will measure the extent to which DNA damage results would be considered trustworthy using a survey.
Extent to which participants believe the feedback to be accurate | Week 3
  The study will measure the extent to which DNA damage results would be considered accurate using an interview.
Extent to which participants believe the feedback to be trustworthy | Week 3
  The study will measure the extent to which DNA damage results would be considered trustworthy using an interview.

SECONDARY OUTCOMES:
Effect size of the changes in coherence between the control and biomarker arm from baseline to three months post-intervention on | Baseline to 3 months
  Change in coherence, as measured by likert scale
Effect size of the change in risk appraisals between the control and biomarker arm from baseline to three months post-intervention on | Baseline to 3 months
  Change in risk appraisals, as measured by a scale
Effect size of participant motivation to quit smoking between the control and biomarker arm from baseline to three months post-intervention on | Baseline to 3 months
  Change in motivation to quit, as measured by a motivation to quit scale
Effect size of plans to quit smoking between the control and biomarker arm from baseline to three months post-intervention on | Baseline to 3 months
  Change in action planning, as measured by number of participants who have made a plan to quit smoking
Effect size of mean levels of smoking between the control and biomarker arm at three months post-intervention | 3 months
  Mean levels of smoking at 3 months
Effect size of the number of quit attempts between the control and biomarker arm at three months post-intervention | 3 months
  Number of quit attempts at 3 months
Effect size of the quit rate between the control and biomarker arm at three months post-intervention | 3 months
  Quit rate at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No